CLINICAL TRIAL: NCT02483260
Title: Intravenous Ribavirin Protocol to Treat Individuals With Viral Hemorrhagic Fever (Crimean-Congo Hemorrhagic Fever or Lassa Fever)
Brief Title: Intravenous Ribavirin Protocol to Treat Individuals With Viral Hemorrhagic Fever
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S-13-08
Record Dates: First submitted 2015-06-24; First posted 2015-06-26 (Estimated); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Viral Hemorrhagic Fever
MeSH Terms: conditions — Hemorrhagic Fevers, Viral | interventions — Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 10-day course of treatment (Other): 10-day course of treatment with follow-up 14 ± 2 days after first dose
  Interventions: Drug: Ribavirin

INTERVENTIONS:
Drug: Ribavirin — 1. Loading dose, 33 mg/kg (maximum dose: 2.64 g)
  2. Followed in 6 hours by a dose of 16 mg/kg (maximum dose: 1.28 g) every 6 hours for the first 4 days (15 doses)
  3. Followed by a dose of 8 mg/kg (maximum dose: 0.64 g) every 8 hours for the subsequent 6 days (18 doses).
  Other Names: Virazole

SUMMARY:
Is ribavirin a therapeutic option for patients with a probable or suspected case of viral hemorrhagic fever?

DETAILED DESCRIPTION:
To provide an intravenous ribavirin therapeutic option for patients with a probable or suspected case of viral hemorrhagic fever, specifically Crimean-Congo hemorrhagic fever or Lassa fever.

ELIGIBILITY:
Inclusion Criteria:

* Meets the case definition for a probable or a suspected case of CCHF or LF
* Must be DoD-affiliated personnel including active and reserve component service members, US civilian employees, contractors, other US personnel, and dependents as well as allied military forces and local nationals who have been granted access to the medical facility
* Is at least 18 years of age (17, if active military) and not greater than 65 years of age
* Has a blood sample drawn and a type and cross-match ordered for transfusion
* Has a hemoglobin greater than or equal to10 g/dL before starting IV ribavirin
* Agrees to collection of required specimens
* Agrees to report any adverse events for the duration of the protocol
* Agrees to a follow-up visit and to donate blood and urine specimens at Day 14 (±2 days) after the first dose of IV ribavirin and agrees to all follow-up visits for anemia or other medical conditions as required by the attending physician
* Female patient of childbearing potential must have a pregnancy test. Patient will be counseled concerning the risks of IV ribavirin versus no treatment if the pregnancy test is positive. If the test is negative, patient agrees to take precautions to avoid pregnancy during treatment and for 7 months after treatment.
* Male patient agrees not to have intercourse with a pregnant woman and to take precautions to avoid producing pregnancies during treatment and for 7 months after ribavirin treatment.
* Female patient agrees not to breastfeed during treatment and for 7 months after ribavirin treatment

Exclusion Criteria:

* • Has known intolerance to ribavirin.

  * Is irreversibly ill on presentation, as defined by presence of profound shock (shock which does not respond to supportive therapy within 3 hours after admission).
  * Has hemoglobin less than 10 g/dL that cannot be corrected to 10 g/dL before initiation of IV ribavirin
  * Has history of hemoglobinopathies (ie, sickle-cell anemia or thalassemia major).
  * Has history of autoimmune hepatitis.
  * Has serum calculated creatinine clearance of < 30 mL/min.
  * History of second or third degree heart block or sick sinus syndrome without a pacemaker and no capability of a pacemaker placement or Wolfe-Parkinson-White Syndrome.
  * A sinus bradycardia of less than 40 beats per minute (see below).
  * Is currently being treated with didanosine (ddI). ddI must be discontinued before starting IV ribavirin.

Relative Exclusion Criteria: At the principal investigator's (PI) discretion, an individual may be treated with IV ribavirin, with caution, if one or more of these criteria are present.

* A positive pregnancy test. The patient will be informed of the risk and benefit of treatment with IV ribavirin versus no ribavirin treatment for CCHF (generally associated with high mortality) and severe cases of Lassa fever (high mortality rates) versus mild cases of Lassa fever (low mortality rates).
* A New York Heart Association cardiac functional capacity of Class II or greater for atherosclerotic heart disease (ASHD) and congestive heart failure (CHF).
* Known cardiac defects that may predispose the subject to bradyarrhythmias, such as second or third degree heart block or sick sinus syndrome without a pacemaker, but capability of pacemaker placement, if needed.
* Sinus bradycardia of 41-49 beats per minutes, if the individual is not known to have a low resting heart rate related to physical conditioning.
* Use of drugs known to result in bradyarrhythmias (certain beta blockers and calcium channel blockers, digoxin, as well as clonidine, cholinesterase inhibitors, and lithium).
* History of gout

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-06-16 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Adverse reactions | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Hawley-Molloy, MD, Principal Investigator — Landstahl Regional Medical Center
Locations (1):
- Landstuhl Regional Medical Center, Landstuhl, APO AE, Germany